CLINICAL TRIAL: NCT00726180
Title: Evaluation of the Use of Trastuzumab to Induce Increased ER Expression in ER-Negative/Low, Her-2/Neu Positive Breast Cancer
Brief Title: Use of Trastuzumab to Induce Increased ER Expression in ER-negative/Low, Her-2/Neu Positive Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to low enrollment
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Ann Schott, MD, Associate Professor of Medicine, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.130
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Results first posted 2013-10-15 (Estimated); Last update posted 2013-10-15 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Women; w/Her2; positive; ERnegative; not metastasized
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: trastuzumab (Herceptin®)

INTERVENTIONS:
Drug: trastuzumab (Herceptin®) — About 1 week (4 - 7 days) before scheduled breast surgery, consisting of lumpectomy or mastectomy, subjects will receive a dose of trastuzumab (Herceptin®). Trastuzumab will be given through an IV or port for approximately 90 minutes. During this time, subjects will be closely monitored by a chemotherapy nurse to make sure that subjects do not have a reaction to the medication. It is possible that the infusion of the medication will need to be slowed down, in which case, the time for the infusion will be longer than 90 minutes. The one dose of the trastuzumab drug will be provided by the study (not billed to insurance), but the charges to administer the drug will be billed to subjects or subjects health insurance.

SUMMARY:
The majority pf breast cancers present as ER-positive, many of which are able to be targeted with multiple hormonal therapies. Altering ER-negative tumors to increase ER expression has the potential to benefit patients by making hormonal therapies a therapeutic option and possibly improving their overall prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Women who have Her-2 positive and ER- negative or ER-low breast cancer that has not metastasized, or spread to other parts of the body, are eligible for the study.
* Participants must have had either a core biopsy or incisional biopsy of their breast cancer, but not yet had definitive breast surgery, including lumpectomy or mastectomy.
* Participants may not have had a BRCA mutation found on genetic testing.
* Participants should have not yet received treatment for their breast cancer, including:

  * chemotherapy,
  * hormonal therapy,
  * trastuzumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schott, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: trastuzumab (Herceptin®) : About 1 week (4 - 7 days) before scheduled breast surgery, consisting of lumpectomy or mastectomy, subjects will receive a dose of trastuzumab (Herceptin®). Trastuzumab will be given through an IV or port for approximately 90 minutes. During this time, subjects will be closely monitored by a chemotherapy nurse to make sure that subjects do not have a reaction to the medication. It is possible that the infusion of the medication will need to be slowed down, in which case, the time for the infusion will be longer than 90 minutes. The one dose of the trastuzumab drug will be provided by the study (not billed to insurance), but the charges to administer the drug will be billed to subjects or subjects health insurance.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Standard Immunohistochemistry and Allred Scores Were to be Used to Measure the Estrogen Receptor (ER) Response Rate in Patients With ER-negative/Low, and Human Epidermal Growth Factor Receptor 2 (HER2)/Neu-positive Breast Cancer.
Time Frame: 90 days
Population: Only 1 patient was enrolled to this study, so no data was obtained.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes